CLINICAL TRIAL: NCT03265236
Title: Diagnostic Value of Antibodies Against a Modified Citrullinated Vimentin in Patients With Rheumatoid Arthritis
Brief Title: Diagnostic Value of Anti-MCV in Pts With RA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Jian Hashim Mohammed, Reident doctor, Assiut University
Other Study IDs: diagnostic value of Anti-MCV
Record Dates: First submitted 2017-08-27; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Anti-MCV in Rheamatoid Arthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group1: Patients with early rheamatoid arthritis
  Interventions: Diagnostic Test: Anti - modified citrullinate vimentin
- Group 2: patients with late rheamatoid arthritis
  Interventions: Diagnostic Test: Anti - modified citrullinate vimentin
- Group 3: Healthy control

INTERVENTIONS:
Diagnostic Test: Anti - modified citrullinate vimentin — patients with early and late RA
  Groups: Group 2; Group1

SUMMARY:
The aim of this work is to evaluate the diagnostic value of anti-MCV antibodies in rheamatoid arthritis patients and to correlate its relationtion disease activity and manifestations.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic systemic autoimmune disease characterized by joint inflammation, subsequent joint destruction leading to loss of joint function, and disability. Joint erosions develop quickly in 25 % of RA patients during the first 3 months of the disease and in about 75% of patients during the first 2years .

Early therapeutic intervention with synthetic disease-modifying antirheumatic drugs (sDMARD) and biological agents that target specific molecules can prevent joint damage and improve the prognosis of the disease. Since these therapies can have potential toxic effects ,it is very important that practitioners diagnose early and reliably the disease, especially the more aggressive forms, in order to select the appropriate treatment for patients.

Early diagnosis of RA can be challenging. During the last 15 years, there has been significant progress on the pathogenesis of RA with the discovery of antibodies against citrullinated protein antigens (ACPAs). ACPA production is associated with the HLA-DRB1 shared epitope, cigarette smoking, and periodontitis .

ACPAs have been shown to predict joint damage and are associated with more severe disease and extra-articular manifestations . In order to better identify RA patients at earlier stages, new 2010 classification criteria for RA by the American College of Rheumatology (ACR)/European League against Rheumatism (EULAR) include rheumatoid factor (RF) and ACPAs .

The most common commercial assay for the detection of ACPAs is anti-cyclic citrullinated peptide (anti-CCP) test, which uses synthetic cyclic citrullinated peptides that mimic RA epitopes.

Citrullination occurs also in other autoimmune diseases .

. Indeed, histone citrullination may lead to the release of neutrophil extracellular traps, and juxtaposition of citrullinated histones with infectious pathogens, complement and immune complexes may compromise tolerance of nuclear autoantigens and promote autoimmunity .

Antibodies to other citrullinated peptides or proteins have been suggested as good candidates for diagnosing RA.

Anti-MCV antibodies have been recommended to be better diagnostic marker for early arthritis .

Vimentin is an intermediate filament that is widely expressed by mesenchymal cells and macrophages and easy to detect in the synovium. Modification of the protein occurs in macrophages undergoing apoptosis, and antibodies to citrullinatedvimentin may emerge if the apoptotic material is inadequately cleared .

ELIGIBILITY:
Inclusion Criteria:

* . All patients were previously diagnosedaccording to the 2010 ACR/EULAR RA classification .. with both ( early and late ) rheamatoid arthritis

Exclusion Criteria:

* patients with other autoimmune disease .
* patient with renal diseaes .

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sixty RA patients attendingAssiut university hospital , and 25 healthy controls were involved in this study. All patients were previously diagnosed according to the 2010 ACR/EULAR RA classification criteria
  The patients and control are divided into:
  * Group I: 30 patients with Early RA
  * Group II:30 patients with Late RA
  * Group III: 25 Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2017-09-15 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
positive Anti-MCV in RA patient | 1 day
  early diagnosis of RA patients by Anti-Mcv antibodies

CONTACTS AND LOCATIONS:
Overall Officials: assiut university, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott DL. Radiological progression in established rheumatoid arthritis. J Rheumatol Suppl. 2004 Mar;69:55-65. PMID 15053455
- [Background] Sakkas LI, Bogdanos DP, Katsiari C, Platsoucas CD. Anti-citrullinated peptides as autoantigens in rheumatoid arthritis-relevance to treatment. Autoimmun Rev. 2014 Nov;13(11):1114-20. doi: 10.1016/j.autrev.2014.08.012. Epub 2014 Aug 23. PMID 25182207
- [Background] Syversen SW, Gaarder PI, Goll GL, Odegard S, Haavardsholm EA, Mowinckel P, van der Heijde D, Landewe R, Kvien TK. High anti-cyclic citrullinated peptide levels and an algorithm of four variables predict radiographic progression in patients with rheumatoid arthritis: results from a 10-year longitudinal study. Ann Rheum Dis. 2008 Feb;67(2):212-7. doi: 10.1136/ard.2006.068247. Epub 2007 May 25. PMID 17526555
- [Background] 9. Khalifa IA (2013 ), Lotfy AM, Elsayed MA, Abd-Elfattah A, Ashraf Abdelmonem A . Anti-Mutated CitrullinatedVimentin Antibodies in Rheumatoid Arthritis compared with anti-cyclic citrullinated peptides. J Am Sci 9: 160-166.
- [Background] Muller S, Radic M. Citrullinated Autoantigens: From Diagnostic Markers to Pathogenetic Mechanisms. Clin Rev Allergy Immunol. 2015 Oct;49(2):232-9. doi: 10.1007/s12016-014-8459-2. PMID 25355199
- [Background] Luime JJ, Colin EM, Hazes JM, Lubberts E. Does anti-mutated citrullinated vimentin have additional value as a serological marker in the diagnostic and prognostic investigation of patients with rheumatoid arthritis? A systematic review. Ann Rheum Dis. 2010 Feb;69(2):337-44. doi: 10.1136/ard.2008.103283. Epub 2009 Mar 15. PMID 19289382
- [Background] Pincus T, Summey JA, Soraci SA Jr, Wallston KA, Hummon NP. Assessment of patient satisfaction in activities of daily living using a modified Stanford Health Assessment Questionnaire. Arthritis Rheum. 1983 Nov;26(11):1346-53. doi: 10.1002/art.1780261107. PMID 6639693
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Ann Rheum Dis. 2010 Sep;69(9):1580-8. doi: 10.1136/ard.2010.138461. PMID 20699241